CLINICAL TRIAL: NCT06917079
Title: A Phase 1a/1b Open-Label Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of BBO-11818 in Subjects With Advanced KRAS Mutant Cancers
Brief Title: BBO-11818 in Adult Subjects With KRAS Mutant Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: TheRas, Inc., d/b/a BBOT (BridgeBio Oncology Therapeutics) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TBBO11818-101; KONQUER-101 (Other: TheRas, Inc., d/b/a BBOT (BridgeBio Oncology Therapeutics))
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-08

CONDITIONS: Non-Small Cell Lung Cancer; NSCLC; PDAC - Pancreatic Ductal Adenocarcinoma; CRC (Colorectal Cancer); Metastatic Non-Small Lung Cell Cancer; Metastatic Colorectal Cancer (CRC); KRAS G12A; KRAS G12C; KRAS G12D; KRAS G12S; KRAS G12V; Metastatic Pancreatic Ductal Adenocarcinoma; Advanced Lung Carcinoma; Solid Tumor, Adult
Keywords: BBOT; BridgeBio Oncology Therapeutics; Phase1; Phase 1a/1b; NSCLC; CRC; PDAC; Metastatic Cancer; Advanced Cancer; Pembrolizumab; Cetuximab; Platinum Chemotherapy; Pemetrexed; KONQUER; KONQUER-101; FOLFOX; NALIRIFOX; Gemcitabine; Nab-paclitaxel
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Neoplasm Metastasis | interventions — pembrolizumab; Cisplatin; Carboplatin; Pemetrexed; Cetuximab; Folfox protocol; Gemcitabine; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Intervention Model Description: Phase 1a: sequential/parallel, Phase 1b: parallel
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (14):
- Cohort 1a - Dose Escalation Monotherapy (Experimental): Participants enrolled in this cohort will receive BBO-11818 as monotherapy
  Interventions: Drug: BBO-11818
- Cohort 1b - Dose Escalation Combination Therapy (Pembrolizumab) (Experimental): Participants enrolled in this cohort will receive BBO-11818 in combination with pembrolizumab infusion (IV)
  Interventions: Drug: BBO-11818; Drug: Pembrolizumab
- Cohort 1c - Dose Escalation Combination Therapy (Pembrolizumab + Cis/carboplatin + Pemetrexed) (Experimental): Participants enrolled in this cohort will receive BBO-11818 in combination with pembrolizumab infusion (IV), cis/carboplatin infusion (IV), and pemetrexed infusion (IV)
  Interventions: Drug: BBO-11818; Drug: Pembrolizumab; Drug: Platinum chemotherapy (cisplatin or carboplatin); Drug: Pemetrexed
- Cohort 1d - Dose Escalation Combination Therapy (Cetuximab) (Experimental): Participants enrolled in this cohort will receive BBO-11818 in combination with cetuximab infusion (IV)
  Interventions: Drug: BBO-11818; Drug: Cetuximab
- Cohort 1e - Dose Escalation Combination Therapy (FOLFOX + Cetuximab) (Experimental): Participants enrolled in this cohort will receive BBO-11818 in combination with cetuximab infusion (IV) and FOLFOX infusion (IV)
  Interventions: Drug: BBO-11818; Drug: Cetuximab; Drug: FOLFOX
- Cohort 1f - Dose Escalation Combination Therapy (NALIRIFOX) (Experimental): Participants enrolled in this cohort will receive BBO-11818 in combination with NALIRIFOX infusion (IV)
  Interventions: Drug: BBO-11818; Drug: NALIRIFOX
- Cohort 1g - Dose Escalation Combination Therapy (Gemcitabine + Nab-Paclitaxel) (Experimental): Participants enrolled in this cohort will receive BBO-11818 in combination with Gemcitabine infusion (IV) and Nab-Paclitaxel infusion (IV)
  Interventions: Drug: BBO-11818; Drug: Gemcitabine; Drug: Nab-paclitaxel
- Cohort 2a - Dose Expansion Monotherapy (Experimental): Participants enrolled in this cohort will receive BBO-11818 as monotherapy
  Interventions: Drug: BBO-11818
- Cohort 2b - Dose Expansion Combination (Pembrolizumab) (Experimental): Participants enrolled in this cohort will receive BBO-11818 in combination with pembrolizumab infusion (IV)
  Interventions: Drug: BBO-11818; Drug: Pembrolizumab
- Cohort 2c - Dose Expansion Combination Therapy (Pembrolizumab + Cis/carboplatin + Pemetrexed) (Experimental): Participants enrolled in this cohort will receive BBO-11818 in combination with pembrolizumab infusion (IV), cis/carboplatin infusion (IV), and pemetrexed infusion (IV)
  Interventions: Drug: BBO-11818; Drug: Pembrolizumab; Drug: Platinum chemotherapy (cisplatin or carboplatin); Drug: Pemetrexed
- Cohort 2d - Dose Expansion Combination Therapy (Cetuximab) (Experimental): Participants enrolled in this cohort will receive BBO-11818 in combination with cetuximab infusion (IV)
  Interventions: Drug: BBO-11818; Drug: Cetuximab
- Cohort 2e - Dose Expansion Combination Therapy (FOLFOX + Cetuximab) (Experimental): Participants enrolled in this cohort will receive BBO-11818 in combination with cetuximab infusion (IV) and FOLFOX infusion (IV)
  Interventions: Drug: BBO-11818; Drug: Cetuximab; Drug: FOLFOX
- Cohort 2f - Dose Expansion Combination Therapy (NALIRIFOX) (Experimental): Participants enrolled in this cohort will receive BBO-11818 in combination with NALIRIFOX infusion (IV)
  Interventions: Drug: BBO-11818; Drug: NALIRIFOX
- Cohort 2g - Dose Expansion Combination Therapy (Gemcitabine + Nab-Paclitaxel) (Experimental): Participants enrolled in this cohort will receive BBO-11818 in combination with Gemcitabine infusion (IV) and Nab-Paclitaxel infusion (IV)
  Interventions: Drug: BBO-11818; Drug: Gemcitabine; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: BBO-11818 — Participants will receive assigned dose of BBO-11818 orally (PO)
Drug: Pembrolizumab — Patients will receive IV pembrolizumab
  Arms: Cohort 1b - Dose Escalation Combination Therapy (Pembrolizumab); Cohort 1c - Dose Escalation Combination Therapy (Pembrolizumab + Cis/carboplatin + Pemetrexed); Cohort 2b - Dose Expansion Combination (Pembrolizumab); Cohort 2c - Dose Expansion Combination Therapy (Pembrolizumab + Cis/carboplatin + Pemetrexed)
Drug: Platinum chemotherapy (cisplatin or carboplatin) — Patients will receive IV platinum chemotherapy (cisplatin or carboplatin)
  Arms: Cohort 1c - Dose Escalation Combination Therapy (Pembrolizumab + Cis/carboplatin + Pemetrexed); Cohort 2c - Dose Expansion Combination Therapy (Pembrolizumab + Cis/carboplatin + Pemetrexed)
Drug: Pemetrexed — Patients will receive IV pemetrexed
  Arms: Cohort 1c - Dose Escalation Combination Therapy (Pembrolizumab + Cis/carboplatin + Pemetrexed); Cohort 2c - Dose Expansion Combination Therapy (Pembrolizumab + Cis/carboplatin + Pemetrexed)
Drug: Cetuximab — Patients will receive IV cetuximab
  Arms: Cohort 1d - Dose Escalation Combination Therapy (Cetuximab); Cohort 1e - Dose Escalation Combination Therapy (FOLFOX + Cetuximab); Cohort 2d - Dose Expansion Combination Therapy (Cetuximab); Cohort 2e - Dose Expansion Combination Therapy (FOLFOX + Cetuximab)
Drug: FOLFOX — Patients will receive IV FOLFOX
  Arms: Cohort 1e - Dose Escalation Combination Therapy (FOLFOX + Cetuximab); Cohort 2e - Dose Expansion Combination Therapy (FOLFOX + Cetuximab)
Drug: NALIRIFOX — Patients will receive IV NALIRIFOX
  Arms: Cohort 1f - Dose Escalation Combination Therapy (NALIRIFOX); Cohort 2f - Dose Expansion Combination Therapy (NALIRIFOX)
Drug: Gemcitabine — Patients will receive IV Gemcitabine
  Arms: Cohort 1g - Dose Escalation Combination Therapy (Gemcitabine + Nab-Paclitaxel); Cohort 2g - Dose Expansion Combination Therapy (Gemcitabine + Nab-Paclitaxel)
Drug: Nab-paclitaxel — Patients will receive IV Nab-Paclitaxel
  Arms: Cohort 1g - Dose Escalation Combination Therapy (Gemcitabine + Nab-Paclitaxel); Cohort 2g - Dose Expansion Combination Therapy (Gemcitabine + Nab-Paclitaxel)

SUMMARY:
A first in human study to evaluate the safety and preliminary antitumor activity of BBO-11818, a pan-KRAS inhibitor, in subjects with locally advanced unresectable or metastatic KRAS mutant solid tumors.

DETAILED DESCRIPTION:
This is an open-label, multi-center, Phase 1 study designed to evaluate the safety, tolerability, pharmacokinetics, and efficacy of BBO-11818, a pan-KRAS inhibitor, alone and in combination with pembrolizumab, pembrolizumab +/- cis/carboplatin + pemetrexed, cetuximab +/- FOLFOX, NALIRIFOX, or Gemcitabine + Nab-paclitaxel in subjects with locally advanced unresectable or metastatic KRAS mutant solid tumors. The study includes dose escalation phase and dose expansion phase.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented locally advanced and unresectable or metastatic NSCLC, PDAC, CRC, or other solid tumor with KRAS G12A, G12C, G12D, G12S, or G12V mutation
* Measurable disease by RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1

Exclusion Criteria:

* Malignancy within the last 2 years as specified in the protocol
* Untreated brain metastases
* Known hypersensitivity to BBO-11818 or its excipients

Other inclusion/exclusion criteria are specified in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 387 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment emergent adverse events (TEAEs), serious adverse events (SAEs), and dose-limiting toxicities (DLTs) | approximately 5 years
Determine recommended dose of BBO-11818 in combination with pembrolizumab +/- cis/carboplatin + pemetrexed, or cetuximab +/- FOLFOX, NALIRIFOX, or Gemcitabine + Nab-paclitaxel | approximately 5 years

SECONDARY OUTCOMES:
Objective response rate (ORR) per RECIST v1.1 and CNS RECIST | approximately 5 years
Clinical benefit rate (CBR) per RECIST v1.1 | approximately 5 years
Duration of Response (DOR) per RECIST v1.1 | approximately 5 years
Progression-Free Survival (PFS) per RECIST v1.1 | approximately 5 years
Overall Survival (OS) | approximately 5 years
Pharmacokinetics of BBO-11818, irinotecan, and SN-38: Maximum blood concentration (Cmax) | approximately 5 years
Pharmacokinetics of BBO-11818, irinotecan, and SN-38: Time to achieve Cmax (Tmax) | approximately 5 years
Pharmacokinetics of BBO-11818, irinotecan, and SN-38: Area under the concentration-time curve (AUC) | approximately 5 years

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - University of California San Diego Moores Cancer Center, San Diego, California
  - Moffitt Cancer Center, Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - NYU Langone Health, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Sarah Cannon Research Institute at Mary Crowley, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah